CLINICAL TRIAL: NCT04302129
Title: ERECTOR SPINAE PLANE BLOCK COMBINED WITH GENERAL ANAESTHESIA VERSUS CONVENTIONAL GENERAL ANAESTHESIA IN LUMBAR SPINE SURGERY
Brief Title: Ultrasound Guided Erector Spinae Plane Block Combined With General Anaesthesia Versus Conventional General Anaesthesia in Lumbar Spine Surgery
Acronym: US ESP block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mohamed Elsayed (Other)
Collaborators: University of Alexandria (Other)
Responsible Party: Sponsor-Investigator, Mohamed Elsayed, doctor, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: operative lumbar spine pain
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Anaesthetic Drugs, Hypotensive Drugs, Perioperative Analgesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: closed envelope method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound guided erector spinae block and general anaesthesia (Experimental): Ultrasound guided erector spine plane block is done after general anaesthesia and prone positioning
  Interventions: Procedure: Erector spinae plane block
- Multimodal analgesia with general anaesthesia (Active Comparator): Multimodal analgesia given with general anaesthesia in form of ketorolac and paracetamol
  Interventions: Drug: Multimodal analgesia

INTERVENTIONS:
Procedure: Erector spinae plane block — 20 ml local anaesthetic are injected bilaterally on each side of the surgical incision underneath the erector spinae muscle where the dorsal rami pass around the bases of the transverse processes.
  Arms: ultrasound guided erector spinae block and general anaesthesia
Drug: Multimodal analgesia — Ketorolac 0.75 mg/ Kg and paracetamol 10 mg/ Kg intravenously
  Arms: Multimodal analgesia with general anaesthesia

SUMMARY:
Ultrasound guided erector spinae plain block combined with general anaesthesia versus conventional general anaesthesia in lumbar spine surgery, it's hypothesized that combined regional anaesthesia with general anaesthesia in lumbar spine surgery may reduce the anaesthetic requirements, aid in controlled hypotension and improve the perioperative pain management.

DETAILED DESCRIPTION:
Primary outcomes:

• Anaesthetic requirements: based on entropy monitoring(state and response entropy monitoring and the difference as a measure for adequacy of analgesia) and haemodynamic parameters ( heart rate and mean arterial blood pressure) at the following time intervals: before induction, after induction, after giving either ESP block or multimodal analgesia and starting surgical stimulus, at 30 min intervals, at end of anaesthesia, at eye opening.

Secondary outcomes:

* Stress response measurement based on serum cortisol and blood glucose levels
* Controlled hypotensive anaesthesia: various drugs required and doses given
* Intraoperative and postoperative analgesia.
* Postanaesthesia care unit data concerning recovery.

ELIGIBILITY:
Inclusion Criteria:

patients undergoing lumbar spine surgery

Exclusion Criteria:

* Coagulation disorders.
* BMI > 30 or < 18.5.
* Patients with surgical site infection.
* Patients with unstable spine integrity like fractures or scoliosis.
* Hypertensive ,cardiac and diabetic patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-04 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Anaesthetic requirements: | the surgery period
  based on entropy monitoring and haemodynamic parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria faculty of medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: After May 2020
Access Criteria: Anaesthetic requirements, Haemodynamic parameters, entropy monitoring, perioperative pain evaluation